CLINICAL TRIAL: NCT00893789
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dosage Study to Evaluate the Efficacy and Safety of Armodafinil (50, 150, and 250 mg/Day) as Treatment for Patients With Excessive Sleepiness Associated With Mild or Moderate Closed Traumatic Brain Injury
Brief Title: Study to Evaluate the Efficacy and Safety of Armodafinil as Treatment for Patients With Excessive Sleepiness Associated With Mild or Moderate Closed Traumatic Brain Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been stopped by sponsor decision.
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/3067/ES/MN
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): Armodafinil 50 mg/day
  Interventions: Drug: Armodafinil
- 2 (Experimental): Armodafinil 150 mg/day
  Interventions: Drug: Armodafinil
- 3 (Experimental): Armodafinil 250 mg/day
  Interventions: Drug: Armodafinil
- 4 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Armodafinil — Armodafinil 50 mg/day
  Arms: 1
Drug: Armodafinil — Armodafinil 150 mg/day
  Arms: 2
Drug: Armodafinil — Armodafinil 250 mg/day
  Arms: 3
Other: Placebo — Placebo
  Arms: 4

SUMMARY:
The primary objective of the study is to determine whether armodafinil treatment is more effective than placebo treatment in patients with excessive sleepiness associated with mild or moderate closed traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

* The patient had a mild (Glasgow Coma Scale [GCS] score 13-15) or moderate (GCS score 9-12) closed TBI at the time of the injury, and the injury occurred 1 to 10 years prior to screening.
* The patient had a Glasgow Outcome Scale score of 5 at the screening visit.
* The patient had an Epworth Sleepiness Scale (ESS) score of at least 10 at screening.
* The patient had a mean sleep latency on the Multiple Sleep Latency Test (MSLT) (average of 4 naps) of less than 8 minutes at baseline.
* The patient had a Clinical Global Impression of Severity of Illness (CGI-S) rating relating to their excessive sleepiness of 4 or more at the screening and baseline visits.
* The patient had a complaint of excessive sleepiness (at least 5 days/week on average) for at least 3 months, and the excessive sleepiness began within 12 months of the TBI.
* Written informed consent was obtained.
* The patient was a man or woman of any ethnic origin 18 to 65 years of age.
* If admitted to an inpatient treatment facility, the patient was discharged at least 1 month prior to the screening visit.
* The patient did not have any medical or psychiatric disorders that could account for the excessive sleepiness.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), used a medically accepted method of contraception, and continued use of one of these methods for the duration of the study (and for 30 days after participation in the study). Acceptable methods of contraception included: abstinence, barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method, or intrauterine device (IUD).
* The patient was in otherwise good health, as judged by the investigator, on the basis of a medical and psychiatric history, physical examination, electrocardiogram (ECG), serum chemistry, hematology, and urinalysis.
* The patient was willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.
* The patient had a Mini Mental State Examination (MMSE) score of more than 26 at the screening visit.
* The patient was on stable dosages of medications (allowed by the protocol) for a minimum of 3 months (selective serotonin reuptake inhibitors [SSRIs] and serotonin-norepinephrine reuptake inhibitors [SNRIs]), 8 weeks (contraceptives), or 4 weeks (all other allowed medication) before the screening visit and was not likely to require a change in therapy for at least 12 weeks on the basis of the investigators' assessment.
* The patient had a habitual bedtime between 2100 and 2400.
* The patient had no other head injuries that, based on medical record documentation or history from the patient and reliable informant (if available), were temporally related to the onset or to any worsening of excessive sleepiness.
* The patient had no other head injury fulfilling the criteria for TBI within ±1 year of the TBI identified according to criterion (a1).

Exclusion Criteria:

* The patient had a history of 2 or more episodes of transient loss of consciousness (LOC) without clear medical explanation, or had a history of known or suspected pseudo seizure (psychogenic seizure). Patients with a history of seizure or epilepsy may have been eligible following discussion with the medical monitor.
* The patient required, or was likely to require, treatment with anticonvulsant medication during the study, or had taken anticonvulsant medication within 6 months before the screening visit.
* The patient had an unstable or uncontrolled medical (including illnesses related to the cardiovascular [including patients with a history of left ventricular hypertrophy or in patients with mitral valve prolapse who had experienced the mitral valve prolapse syndrome], renal, or hepatic systems or surgical) condition (treated or untreated) or was not a suitable candidate for treatment with armodafinil, as judged by the investigator.
* The patient had neurosurgery involving the brain or brainstem.
* The patient had a history of schizophrenia, bipolar disorder, psychotic depression, or other psychotic episode.
* The patient had any current Axis I disorder (including depression and posttraumatic stress disorder [PTSD]), as assessed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (SCID). The patient had any Axis II disorder (as assessed by SCID) that, in the opinion of the investigator, would affect patient participation in the study or full compliance with study procedures.
* The patient had a history of, or currently met The International Classification of Sleep Disorders, Edition 2 (ICSD 2) (American Academy of Sleep Medicine 2005) criteria for narcolepsy, obstructive sleep apnea/hypopnea syndrome (OSAHS), shift work sleep disorder (SWSD), or any other sleep disorder associated with excessive daytime sleepiness; or the patient had a history of idiopathic hypersomnia, insomnia (requiring treatment), or sleep disorder before the development of the TBI.
* The patient had 85% or less sleep efficiency (sleep duration ÷ time in bed x 100%) as determined from nocturnal polysomnography (NPSG).
* The patient had any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The patient used any medications, including over-the-counter (OTC) medicines disallowed by the protocol, within 7 days or 5 half lives (medication or its active metabolites), whichever was longer, before the screening visit.
* The patient had a need for chronic pain medications.
* In the judgment of the investigator, the patient had a clinically significant deviation from normal in the physical examination.
* In the judgment of the investigator, the patient had any clinically significant ECG finding.
* The patient had a diagnosis of any type of dementia.
* The patient had a history of suicidal ideation (considered by the investigator to be of current clinical significance), or was currently suicidal.
* The patient had a known hypersensitivity to armodafinil, racemic modafinil, or any component of the study drug tablets. Armodafinil tablets contain the following inactive ingredients: croscarmellose sodium, lactose, magnesium stearate, microcrystalline cellulose, povidone, and pregelatinized starch.
* The patient had a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions.
* The patient had a clinical laboratory test value(s) outside the range(s) specified by protocol (or any other clinically significant laboratory abnormality), and the medical monitor had not provided written approval for study participation.
* The patient had a history (within the past 5 years) of alcohol, narcotic, or any other drug abuse (with the exception of nicotine) as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition, Text Revision (DSM-IV-TR), or the patient had current evidence of substance use, without medical explanation, confirmed by results of a urine drug screen (UDS).
* The patient had taken armodafinil, modafinil or other stimulant medication for excessive sleepiness within 1 month of the screening visit.
* The patient was a pregnant or lactating woman. (Any women becoming pregnant during the study were to be withdrawn from the study.)
* The patient was known to have tested positive for human immunodeficiency virus (HIV).
* The patient consumed an average of more than 600 mg of caffeine per day, including coffee, tea and/or other caffeine-containing beverages or food.
* The patient used any investigational drug within 1 month before the screening visit.
* The patient was receiving workmen's compensation or was in active litigation with regard to TBI.
* The patient had a self-reported Hamilton Depression Rating Scale, 6 Item Version (S HAM D6) score of more than 4 at the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (73):
- United States (68):
  - Teva Investigational Site 58, Birmingham, Alabama
  - Teva Investigational Site 62, Tucson, Arizona
  - Teva Investigational Site 40, Tucson, Arizona
  - Teva Investigational Site 16, Hot Springs, Arkansas
  - Teva Investigational Site 5, Little Rock, Arkansas
  - Teva Investigational Site 44, Fountain Valley, California
  - Teva Investigational Site 49, La Palma, California
  - Teva Investigational Site 51, La Palma, California
  - Teva Investigational Site 71, Mather, California
  - Teva Investigational Site 55, San Diego, California
  - Teva Investigational Site 33, San Diego, California
  - Teva Investigational Site 53, Santa Monica, California
  - Teva Investigational Site 69, Wallingford, Connecticut
  - Teva Investigational Site 52, Hallandale, Florida
  - Teva Investigational Site 47, Miami, Florida
  - Teva Investigational Site 1, Orlando, Florida
  - Teva Investigational Site 18, Pembroke Pines, Florida
  - Teva Investigational Site 10, Spring Hill, Florida
  - Teva Investigational Site 38, St. Petersburg, Florida
  - Teva Investigational Site 17, Tampa, Florida
  - Teva Investigational Site 26, Atlanta, Georgia
  - Teva Investigational Site 12, Atlanta, Georgia
  - Teva Investigational Site 14, Atlanta, Georgia
  - Teva Investigational Site 68, Gainesville, Georgia
  - Teva Investigational Site 67, Macon, Georgia
  - Teva Investigational Site 29, Stockbridge, Georgia
  - Teva Investigational Site 15, Suwanee, Georgia
  - Teva Investigational Site 46, Chicago, Illinois
  - Teva Investigational Site 54, Chicago, Illinois
  - Teva Investigational Site 59, Chicago, Illinois
  - Teva Investigational Site 28, Danville, Indiana
  - Teva Investigational Site 19, Fort Wayne, Indiana
  - Teva Investigational Site 2, Indianapolis, Indiana
  - Teva Investigational Site 39, Indianapolis, Indiana
  - Teva Investigational Site 41, Iowa City, Iowa
  - Teva Investigational Site 9, Shawnee Mission, Kansas
  - Teva Investigational Site 48, Louisville, Kentucky
  - Teva Investigational Site 32, Chevy Chase, Maryland
  - Teva Investigational Site 37, Belmont, Massachusetts
  - Teva Investigational Site 70, Brighton, Massachusetts
  - Teva Investigational Site 22, Saginaw, Michigan
  - Teva Investigational Site 7, Hattiesburg, Mississippi
  - Teva Investigational Site 42, St Louis, Missouri
  - Teva Investigational Site 56, Lincoln, Nebraska
  - Teva Investigational Site 72, New York, New York
  - Teva Investigational Site 63, New York, New York
  - Teva Investigational Site 36, West Seneca, New York
  - Teva Investigational Site 11, Durham, North Carolina
  - Teva Investigational Site 45, Winston-Salem, North Carolina
  - Teva Investigational Site 31, Cincinnati, Ohio
  - Teva Investigational Site 34, Cincinnati, Ohio
  - Teva Investigational Site 57, Middleburg Heights, Ohio
  - Teva Investigational Site 30, Toledo, Ohio
  - Teva Investigational Site 3, Oklahoma City, Oklahoma
  - Teva Investigational Site 64, Clarks Summit, Pennsylvania
  - Teva Investigational Site 13, Jefferson Hills, Pennsylvania
  - Teva Investigational Site 65, Columbia, South Carolina
  - Teva Investigational Site 61, Germantown, Tennessee
  - Teva Investigational Site 60, Austin, Texas
  - Teva Investigational Site 25, Dallas, Texas
  - Teva Investigational Site 8, Houston, Texas
  - Teva Investigational Site 20, Houston, Texas
  - Teva Investigational Site 73, Kingwood, Texas
  - Teva Investigational Site 23, San Antonio, Texas
  - Teva Investigational Site 35, Midvale, Utah
  - Teva Investigational Site 66, Midvale, Utah
  - Teva Investigational Site 24, Richmond, Virginia
  - Teva Investigational Site 50, West Allis, Wisconsin
- Germany (2):
  - Teva Investigational Site 405, Berlin
  - Teva Investigational Site 404, München
- Teva Investigational Site 501, Pisa, Italy
- Spain (2):
  - Teva Investigational Site 704, Barcelona
  - Teva Investigational Site 701, Madrid

REFERENCES:
- [Derived] Menn SJ, Yang R, Lankford A. Armodafinil for the treatment of excessive sleepiness associated with mild or moderate closed traumatic brain injury: a 12-week, randomized, double-blind study followed by a 12-month open-label extension. J Clin Sleep Med. 2014 Nov 15;10(11):1181-91. doi: 10.5664/jcsm.4196. PMID 25325609

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral placebo tablets, once daily (QD)
- Armodafinil 50 mg/Day: Oral armodafinil 50 mg tablets, once daily (QD)
- Armodafinil 150 mg/Day: Oral armodafinil 150 mg tablets, once daily (QD)
- Armodafinil 250 mg/Day: Oral armodafinil 250 mg tablets, once daily (QD)
Period: Overall Study
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Started | 29 | 30 | 29 | 29
Safety Analysis Set (SAS) | 29 (SAS = all participants who received 1 or more doses of study drug.) | 30 | 29 | 29
Full Analysis Set (FAS) | 29 (FAS = participants in the safety analysis set with ≥1 postbaseline primary efficacy assessment.) | 29 | 28 | 27
Completed | 23 | 26 | 22 | 16
Not Completed | 6 | 4 | 7 | 13
Not completed — Withdrawal by Subject | 3 | 1 | 3 | 1
Not completed — Noncompliance With Study Drug | 1 | 0 | 1 | 2
Not completed — Noncompliance With Study Procedures | 1 | 0 | 0 | 0
Not completed — Taking Excluded Concomitant Medication | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 5
Not completed — Protocol Violation | 0 | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day | Total
Number analyzed (Participants) | 29 | 30 | 29 | 29 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (11.02) | 33.2 (9.31) | 32.3 (10.81) | 29.4 (11.07) | 31.3 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 13 | 53
  Male | 15 | 17 | 16 | 16 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 2
  Black or African American | 2 | 2 | 6 | 4 | 14
  White | 26 | 27 | 22 | 24 | 99
  More than one race | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Multiple Sleep Latency Test (MSLT) at Endpoint (Last Postbaseline Observation Up to Week 12)
Description: The MSLT is an objective assessment of sleepiness that measures the likelihood of falling asleep. Four 20-minute (maximum) MSLT naps were performed at 0900, 1100, 1300, and 1500. The participant, dressed in nonconstricting clothes, was instructed to lie quietly and attempt sleep. Each MSLT nap continued until: (a) 3 consecutive 30-second epochs of stage 1 sleep were reached or (b) any single, 30-second epoch of stage 2, 3, 4, or rapid eye movement (REM) sleep was reached. Sleep latency for each nap and average sleep latency for the 4 naps were tabulated. According to clinical protocol for the MSLT, each nap was terminated after 20 minutes if no sleep occurred. If a participant did not fall asleep in 20 minutes, his/her sleep latency for that nap was set to 20 minutes. Sleep latency was measured as the elapsed time from lights-out to the first epoch scored as sleep. With a 30-second scoring epoch, this criterion was reached when sleep occupied at least 16 seconds of any epoch.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Full Analysis Set (all participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment); n=number of participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 29 | 28 | 27
minutes
  Baseline (BL; n=29, 29, 28, 27) | 3.3 (1.79) | 4.2 (1.69) | 4.2 (2.05) | 3.7 (2.04)
  Change from BL at Endpoint (n=27, 29, 26, 21) | 2.4 (4.03) | 2.6 (4.35) | 5.0 (4.95) | 7.2 (6.35)
Statistical Analysis 1: Comparison: Placebo vs Armodafinil 50 mg/Day; P-value for "Change from Baseline at Endpoint."; Test type: Superiority or Other; p = 0.8336, ANCOVA — The analyses performed were not done in accordance to the study protocol as the study was terminated early and therefore the analyses done were underpowered, no adjustments for multiple comparisons (or step-down analysis rules) were applied
Statistical Analysis 2: Comparison: Placebo vs Armodafinil 150 mg/Day; P-value for "Change from Baseline at Endpoint."; Test type: Superiority or Other; p = 0.0514, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Armodafinil 250 mg/Day; P-value for "Change from Baseline at Endpoint."; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Responders and Nonresponders According to Clinical Global Impression of Change (CGI-C) Ratings at Endpoint (Last Postbaseline Observation Up to Week 12)
Description: The CGI-C is the clinician's rating of disease severity as compared with pretreatment, assessed by the Clinical Global Impression of Severity (CGI-S). Severity of illness, as related to excessive sleepiness, was assessed at baseline by the CGI-S, which consists of 7 categories: normal-shows no sign of illness, borderline ill, mildly (slightly) ill, moderately ill, markedly ill, severely ill, and among the most extremely ill. The clinician assessed the change from baseline in the participant's condition, as related to excessive sleepiness, in response to treatment. The CGI-C uses the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse. Responders were defined as those participants who were considered much or very much improved on the CGI-C. Those in all other categories of the CGI-C were considered nonresponders.
Time Frame: Last postbaseline observation up to Week 12
Population: Full Analysis Set (all participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 29 | 28 | 27
percentage of participants
  Responders | 38 | 41 | 54 | 48
  Nonresponders | 62 | 59 | 46 | 52
Statistical Analysis 1: Comparison: Placebo vs Armodafinil 50 mg/Day; Test type: Superiority or Other; p = 0.7884, Pearson's chi-squared
Statistical Analysis 2: Comparison: Placebo vs Armodafinil 150 mg/Day; Test type: Superiority or Other; p = 0.2359, Pearson's chi-squared
Statistical Analysis 3: Comparison: Placebo vs Armodafinil 250 mg/Day; Test type: Superiority or Other; p = 0.4401, Pearson's chi-squared

3. Secondary Outcome: Change From Baseline in Mean Sleep Latency From the MSLT at Weeks 4, 8, and 12
Description: The MSLT is an objective assessment of sleepiness that measures the likelihood of falling asleep. Four 20-minute (maximum) MSLT naps were performed at 0900, 1100, 1300, and 1500. The participant, dressed in nonconstricting clothes, was instructed to lie quietly and attempt sleep. Each MSLT nap continued until: (a) 3 consecutive 30-second epochs of stage 1 sleep were reached or (b) any single, 30-second epoch of stage 2, 3, 4, or rapid eye movement (REM) sleep was reached. Sleep latency for each nap and average sleep latency for the 4 naps were tabulated. According to clinical protocol for the MSLT, each nap was terminated after 20 minutes if no sleep occurred. Sleep latency was measured as the elapsed time from lights-out to the first epoch scored as sleep. With a 30-second scoring epoch, this criterion was reached when sleep occupied at least 16 seconds of any epoch.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: Full Analysis Set (all participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment); n=number of participants with data at given time points.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 29 | 28 | 27
minutes
  Baseline (BL; n=29, 29, 28, 27) | 3.3 (1.79) | 4.2 (1.69) | 4.2 (2.05) | 3.7 (2.04)
  Change from BL at Week 4 (n=26, 29, 26, 20) | 3.2 (4.93) | 2.7 (5.21) | 4.0 (5.43) | 7.0 (4.80)
  Change from BL at Week 8 (n=24, 27, 24, 17) | 2.1 (4.73) | 2.5 (4.88) | 4.2 (5.94) | 4.2 (5.47)
  Change from BL at Week 12 (n=22, 26, 22, 15) | 1.8 (3.87) | 2.7 (4.53) | 4.6 (4.39) | 7.4 (6.38)

4. Secondary Outcome: Percentage of Responders and Nonresponders According to Clinical Global Impression of Change (CGI-C) Ratings at Weeks 2, 4, 8, and 12
Description: as for outcome 2
Time Frame: Weeks 2, 4, 8, and 12
Population: Full Analysis Set (all participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment); n=number of participants with a nonmissing value at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 29 | 28 | 27
percentage of participants
  Week 2 Responders (n=28, 29, 27, 23) | 14 | 21 | 37 | 39
  Week 2 Nonresponders (n=28, 29, 27, 23) | 86 | 79 | 63 | 61
  Week 4 Responders (n=27, 29, 26, 20) | 22 | 24 | 50 | 50
  Week 4 Nonresponders (n=27, 29, 26, 20) | 78 | 76 | 50 | 50
  Week 8 Responders (n=23, 27, 24, 18) | 35 | 48 | 54 | 56
  Week 8 Nonresponders (n=23, 27, 24, 18) | 65 | 52 | 46 | 44
  Week 12 Responders (n=23, 26, 22, 16) | 35 | 42 | 55 | 56
  Week 12 Nonresponders (n=23, 26, 22, 16) | 65 | 58 | 45 | 44

5. Secondary Outcome: Change From Baseline in Traumatic Brain Injury - Work Instability Scale (TBI-WIS) Total Score At Weeks 4, 8, 12 and Endpoint (Last Postbaseline Observation Up to Week 12)
Description: The TBI-WIS is a validated participant-rated instrument for assessing a participant's functional ability after TBI and the functional demands of their job. The assessment consists of 36 questions to which the participant responded with a "true" or "not true" answer. To score the questionnaire, the number of "true" responses is counted: if < 2, the risk is low; 2 to 23, the risk is medium; and >23, the risk is high, for work instability. Score range is 0 (lowest risk for work instability) to 36 (highest risk for work instability).
Time Frame: Weeks 4, 8, 12 and Endpoint (last postbaseline observation up to Week 12)
Population: Participants in the Full Analysis Set (participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment) with a baseline TBI-WIS measurement; n=number of participants with values at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 24 | 24 | 19 | 21
units on a scale
  Baseline (BL; n=24, 24, 19, 21) | 8.5 (6.75) | 9.3 (8.80) | 8.7 (7.55) | 11.6 (10.71)
  Change from BL at Week 4 (n=23, 23, 18, 15) | -2.5 (4.71) | -2.5 (3.72) | -0.5 (3.71) | -2.8 (3.88)
  Change from BL at Week 8 (n=19, 22, 17, 13) | -1.4 (5.52) | -3.5 (4.94) | -2.4 (5.26) | -4.7 (8.89)
  Change from BL at Week 12 (n=19, 21, 17, 12) | -0.9 (6.27) | -3.9 (4.74) | -2.5 (4.32) | -5.0 (6.90)
  Change from BL at Endpoint (n=24, 24, 19, 19) | -2.3 (6.44) | -3.4 (4.60) | -2.5 (4.07) | -2.5 (7.12)

6. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) at Week 12 and Endpoint (Last Postbaseline Observation Up to Week 12)
Description: The patient's evaluation of excessive daytime sleepiness was measured by the ESS. The ESS score is based on responses to questions referring to 8 everyday situations (eg, sitting and reading, talking to someone, being stopped in traffic) and reflects a patient's propensity to fall asleep in those situations. The ESS score is derived from the sum of the values from questions corresponding to the 8 situations. Scores for the ESS range from 0 to 24, with a higher score indicating a greater daytime sleepiness. This test was self-administered.
Time Frame: Baseline, Week 12, Endpoint (last postbaseline observation, up to Week 12)
Population: Full Analysis Set (all participants who received 1 or more doses of study drug with ≥1 postbaseline primary efficacy assessment); n=number of participants with data at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 29 | 28 | 27
units on a scale
  Baseline (BL; n=29, 29, 28, 27) | 14.8 (2.83) | 14.3 (2.61) | 15.1 (2.54) | 16.1 (3.82)
  Change from BL at Week 12 (n=23, 26, 22, 16) | -5.0 (6.12) | -4.6 (5.30) | -6.5 (4.40) | -9.2 (4.90)
  Change from BL at Endpoint (n=27, 28, 26, 23) | -5.1 (5.93) | -4.5 (5.15) | -6.1 (4.52) | -7.0 (5.61)

7. Secondary Outcome: Percentage of Participants Answering "No" to All Questions on the Columbia-Suicide Severity Rating Scale Since Last Visit Version (C-SSRS SLV) at Weeks 2, 4, 8, 12 and Endpoint (Last Postbaseline Observation Up to Week 12)
Description: The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors since last visit (SLV). The number of participants answering 'no' to all 9 yes/no questions about suicidal behaviors, ideations, and acts are presented. Questions included the presence of the following: a wish to be dead; nonspecific active suicidal thoughts; actual suicide attempt; non-suicidal self-injurious behavior; interrupted attempt; aborted attempt; suicidal behavior; preparatory suicidal acts or behavior; and completed suicide.
Time Frame: Weeks 4, 8, 12 and Endpoint (last postbaseline observation up to Week 12)
Population: Safety analysis set (all participants who received 1 or more doses of study drug); n=all participants with a nonmissing value at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 29 | 29
percentage of participants
  Week 2 (n=14, 14, 13, 12) | 100 | 100 | 100 | 100
  Week 4 (n=13, 16, 15, 11) | 100 | 100 | 100 | 100
  Week 8 (n=13, 15, 13, 10) | 100 | 100 | 100 | 100
  Week 12 (n=14, 15, 13, 9) | 100 | 100 | 100 | 100
  Endpoint (n=19, 18, 16, 15) | 100 | 100 | 100 | 100

8. Secondary Outcome: Change From Baseline in the Total Score From the Self-Reported Hamilton Depression Rating Scale, 6 Item Version (S-HAM-D6) at Weeks 2, 4, 8, 12 and Endpoint (Last Postbaseline Observation Up to 12 Weeks)
Description: The self-reported S-HAM-D6 is a validated scale developed from the core depressive items of the 17 Item Hamilton Depression Inventory (HAM-D17). The HAM-D6 (Items 1, 2, 7, 8, 10, 13 from the 17-item HAMD) evaluates "core" symptoms of Major Depressive Disorder (MDD). The assessment consists of 6 items representing depressed mood, guilt, work and activities, retardation, psychic anxiety, and general somatic symptoms. Each item is evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). Total scores range from 0 (normal) to 22 (severe). Scores greater than 12 indicate moderate to severe depression and scores less than 12 indicate mild depression.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and Endpoint (last postbaseline observation up to 12 weeks)
Population: Participants in the Safety Analysis Set (participants who received 1 or more doses of study drug) with a baseline S-HAM-D6 measurement; n=number of participants with nonmissing data at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 13 | 13 | 11 | 13
units on a scale
  Baseline (BL; n=13, 13, 11, 13) | 1.3 (1.49) | 1.8 (1.07) | 1.2 (1.72) | 1.5 (1.33)
  Change from BL at Week 2 (n=13, 13, 11, 11) | -0.7 (1.38) | -0.5 (2.63) | 0.3 (1.49) | 0.4 (1.29)
  Change from BL at Week 4 (n=12, 12, 11, 10) | -0.5 (1.62) | 0.9 (2.68) | -0.2 (1.47) | 0.2 (2.97)
  Change from BL at Week 8 (n=10, 11, 10, 9) | 0.1 (1.60) | 1.1 (4.68) | -0.2 (1.40) | 1.6 (3.05)
  Change from BL at Week 12 (n=9, 10, 9, 8) | 0.9 (2.80) | 0.2 (2.74) | 1.0 (2.65) | -0.1 (2.17)
  Change from BL at Endpoint (n=13, 13, 11, 13) | 0.5 (2.54) | -0.1 (2.43) | 0.6 (2.54) | 0.9 (4.41)

9. Secondary Outcome: Change From Baseline in the Total Sleep Time As Assessed by Nocturnal Polysomnography (NPSG) at Weeks 2, 4, 12 and Endpoint (Last Postbaseline Observation Up to 12 Weeks)
Description: NPSG continuously records normal and abnormal physiological activity during an entire night. It documents the adequacy of sleep, including the frequency, duration, and total amounts of stage 1-2, stage 3-4 (slow wave sleep), and rapid eye movement (REM) sleep.
Time Frame: Baseline, Weeks 2, 4, 12, and Endpoint (last postbaseline observation up to 12 weeks)
Population: Safety Analysis Set (all participants who received 1 or more doses of study drug); n=number of participants with data at given time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 29 | 29
minutes
  Baseline (BL; n=29, 30, 29, 29) | 442.3 (19.60) | 442.4 (18.38) | 442.0 (19.07) | 442.8 (19.16)
  Change from BL at Week 2 (n=28, 29, 27, 24) | -4.4 (29.62) | 5.8 (27.14) | -3.9 (38.10) | -8.8 (41.85)
  Change from BL at Week 4 (n=26, 28, 26, 21) | -16.9 (78.81) | 2.9 (34.50) | 4.0 (41.32) | -21.6 (51.18)
  Change from BL at Week 12 (n=22, 26, 22, 15) | -0.5 (24.39) | 8.3 (20.46) | -18.3 (62.26) | -33.1 (55.65)
  Change from BL at Endpoint (n=29, 30, 27, 26) | -10.1 (35.75) | 6.6 (21.37) | -19.7 (60.53) | -21.2 (46.77)

10. Secondary Outcome: Plasma Concentrations of Selective Serotonin Reuptake Inhibitors (SSRIs) and Serotonin and Norepinephrine Reuptake Inhibitors (SNRIs) at Weeks 4, 8, and 12 (or Last Postbaseline Observation Up to Week 12)
Description: To evaluate the impact of treatment with armodafinil on the pharmacokinetics of selective serotonin reuptake inhibitors (SSRIs) and serotonin and norepinephrine reuptake inhibitors (SNRIs) (as appropriate), plasma concentrations at weeks 4, 8, and 12 (or last postbaseline observation) were to be assessed.
Time Frame: Weeks 4, 8, and 12 (or last postbaseline observation, up to Week 12)
Population: Due to the limited samples available for measurement of concentrations of antidepressants in the study, the plasma concentrations of antidepressants were not measured. The planned pharmacokinetic evaluation of the impact of armodafinil treatment on the pharmacokinetics of selective antidepressants was not conducted.
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Concomitant Medication Usage In ≥5% of Participants Throughout the Study
Description: Therapeutic classification of concomitant medications used by ≥5% of participants throughout the study. Participants are counted only once in each therapeutic class category. Medications were included in the table if the proportion of participants in the combined armodafinil treatment group was ≥5%.
Time Frame: Screening through Week 12
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 29 | 29
participants
  Analgesics | 4 | 4 | 7 | 6
  Antibacterials | 2 | 2 | 1 | 2
  Antihistamines for systemic use | 1 | 2 | 4 | 2
  Anti-inflammatory and antirheumatic products | 8 | 9 | 5 | 8
  Drugs for acid-related disorders | 0 | 2 | 2 | 2
  Lipid-modifying agents | 2 | 8 | 2 | 2
  Nasal preparations | 2 | 3 | 1 | 2
  Sex hormones and modulators of the genital system | 3 | 4 | 3 | 3
  Unspecified herbal | 1 | 3 | 1 | 1
  Vitamins/nutritional supplement | 5 | 7 | 4 | 7

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Withdrawals Due to AEs
Description: AE=any untoward medical occurrence in a patient that develops or worsens in severity during the conduct of the clinical study of a pharmaceutical product and does not necessarily have a causal relationship to the study drug. SAE=any AE that resulted in any of the following: death; a life-threatening adverse event; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly or birth defect; an important medical event that required medical intervention to prevent 1 of the outcomes listed in this definition. Treatment-related AEs=definite, probable, possible, or missing relationship. Protocol-defined AEs=treatment-emergent adverse events associated with skin rash, hypersensitivity reaction, emergent suicidal ideation or suicide attempt, depression, psychosis (including hypomanic or manic episode), and seizure or suspected seizure were considered to be of potential clinical importance.
Time Frame: Screening through Week 12
Population: Safety Analysis Set (all participants who received 1 or more doses of study drug).
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 29 | 29
participants
  Any adverse event | 14 | 15 | 16 | 16
  Severe adverse events | 0 | 0 | 0 | 0
  Treatment-related adverse events | 8 | 9 | 14 | 15
  Deaths | 0 | 0 | 0 | 0
  Other serious adverse events | 0 | 0 | 0 | 0
  Withdrawn from study due to adverse events | 0 | 2 | 1 | 5
  Protocol-defined adverse event | 0 | 1 | 0 | 3

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Postbaseline Serum Chemistry Values
Description: Normal ranges for serum chemistry values: blood urea nitrogen (BUN), 1.43 - 8.57 mmol/L; uric acid, 124.91 - 493.68 μmol/L; aspartate aminotransferase (AST), 11 - 36 U/L; gamma-glutamyl transpeptidase (GGT), 10 - 61 U/L; total bilirubin, 3.42 - 20.52 μmol/L.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 28 | 28
participants
  BUN >=10.71 mmol/L | 1 | 0 | 0 | 0
  Uric acid >=625 (men) or >=506 (women) μmol/L | 0 | 1 | 0 | 0
  AST >=3 x upper limit of normal | 0 | 0 | 1 | 0
  GGT >=3 x upper limit of normal | 0 | 1 | 0 | 0
  Total bilirubin >=34.2 μmol/L | 0 | 1 | 1 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Postbaseline Hematology Values
Description: Normal ranges for hematology values: white blood cell (WBC) count, 3.8 - 10.7 x 10^9/L; absolute neutrophil count (ANC), 1.96 - 7.23 x 10^9/L. Participants may have had more than one clinically significant abnormal value.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 28 | 28
participants
  WBC <=3.0 x 10^9/L | 1 | 1 | 1 | 0
  ANC <=1.0 x 10^9/L | 1 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Postbaseline Urinalysis Values
Description: Participants with at least one clinically significant postbaseline urinalysis abnormality, specifically presented is blood (hemoglobin) in urine >=2 units increase from baseline.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 28 | 28
participants | 2 | 1 | 1 | 1

16. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Sign Values
Description: Criteria for clinically significant abnormal vital signs values: heart rate, ≤50 beats per minute (bpm) and decrease from baseline of ≥15 bpm; sitting systolic blood pressure, ≤90 mm Hg and decrease from baseline of ≥20 mm Hg; sitting diastolic blood pressure, ≤50 mm Hg and decrease from baseline of ≥15 mm Hg.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 28 | 29
participants
  Heart Rate | 0 | 1 | 1 | 0
  Sitting Systolic Blood Pressure | 0 | 1 | 0 | 0
  Sitting Diastolic Blood Pressure | 0 | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With Notable Blood Pressure Values Per World Health Organization Criteria
Description: Criteria for World Health Organization (WHO) notable blood pressure (BP) values: systolic blood pressure, ≥140 mm Hg plus increase of ≥10% from baseline; diastolic blood pressure, ≥90 mm Hg plus increase of ≥10% from baseline.
Time Frame: Baseline, last postbaseline observation up to Week 12
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 28 | 29
participants
  Sitting Systolic Blood Pressure | 0 | 1 | 1 | 2
  Sitting Diastolic Blood Pressure | 0 | 2 | 0 | 2

18. Secondary Outcome: Electrocardiogram (ECG) Findings Shifts From Baseline to Overall
Description: Number of participants with shifts from normal/abnormal 12-lead ECG findings at baseline (BL) to (→) normal/abnormal findings overall are presented. For overall, the worst postbaseline finding (the abnormal finding if there are both normal and abnormal findings) for the participant between baseline and endpoint (defined as last postbaseline observation, up to Week 12) is summarized. Shifts (normal and abnormal) from baseline to overall are summarized using participant counts. Any ECG finding that was judged by the investigator as a clinically meaningful change (worsening) compared to baseline was recorded as an adverse event.
Time Frame: Baseline through Endpoint (last postbaseline observation, up to Week 12)
Population: Participants in the Safety Analysis Set with a baseline and postbaseline measurement are summarized.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 28 | 27 | 27 | 27
participants
  Normal at BL → Normal Overall | 15 | 16 | 14 | 15
  Normal at BL → Abnormal Overall | 1 | 2 | 4 | 1
  Abnormal at BL → Normal Overall | 3 | 3 | 7 | 3
  Abnormal at BL → Abnormal Overall | 9 | 6 | 2 | 8

19. Secondary Outcome: Physical Examination Findings Shifts From Baseline to Endpoint (Last Postbaseline Observation, up to Week 12)
Description: Number of participants with shifts from normal/abnormal physical examination findings at baseline (BL) to (→) normal/abnormal findings at endpoint (EP, defined as last postbaseline observation, up to Week 12). Shifts (normal and abnormal) from baseline to endpoint are summarized using participant counts for each physical examination category. A newly diagnosed finding was defined as being normal or missing at baseline and abnormal at least once during the study. Any physical examination finding that was judged by the investigator as a clinically significant change (worsening) compared to a baseline value was considered an adverse event. HEENT=head, eyes, ears, nose, throat.
Time Frame: Baseline through Endpoint (last postbaseline observation, up to Week 12)
Population: For each category, only participants in the Safety Analysis Set with a baseline and postbaseline measurement are summarized.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Number analyzed (Participants) | 29 | 30 | 29 | 29
participants
  General Appearance: Normal at BL → Normal at EP | 26 | 27 | 26 | 27
  General Appearance: Normal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  General Appearance: Abnormal at BL → Normal at EP | 0 | 2 | 1 | 0
  General Appearance:Abnormal at BL → Abnormal at EP | 2 | 0 | 0 | 0
  HEENT: Normal at BL→ Normal at EP | 26 | 29 | 24 | 26
  HEENT: Normal at BL→ Abnormal at EP | 1 | 0 | 1 | 0
  HEENT: Abnormal at BL→ Normal at BL | 0 | 0 | 1 | 0
  HEENT: Abnormal at BL→ Abnormal at EP | 1 | 0 | 1 | 1
  Chest/Lungs: Normal at BL→ Normal at EP | 28 | 29 | 27 | 27
  Chest/Lungs: Normal at BL→ Abnormal at EP | 0 | 0 | 0 | 0
  Chest/Lungs: Abnormal at BL→ Normal at EP | 0 | 0 | 0 | 0
  Chest/Lungs: Abnormal at BL→ Abnormal at EP | 0 | 0 | 0 | 0
  Heart: Normal at BL → Normal at EP | 26 | 29 | 27 | 26
  Heart: Normal at BL → Abnormal at EP | 0 | 0 | 0 | 1
  Heart: Abnormal at BL → Normal at EP | 2 | 0 | 0 | 0
  Heart: Abnormal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  Abdomen: Normal at BL → Normal at EP | 27 | 27 | 26 | 26
  Abdomen: Normal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  Abdomen: Abnormal at BL → Normal at EP | 0 | 2 | 1 | 0
  Abdomen: Abnormal at BL → Abnormal at EP | 1 | 0 | 0 | 0
  Musculoskeletal: Normal at BL → Normal at EP | 27 | 29 | 25 | 27
  Musculoskeletal: Normal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  Musculoskeletal: Abnormal at BL → Normal at EP | 1 | 0 | 1 | 0
  Musculoskeletal: Abnormal at BL → Abnormal at EP | 0 | 0 | 1 | 0
  Skin: Normal at BL → Normal at EP | 25 | 24 | 24 | 24
  Skin: Normal at BL → Abnormal at EP | 0 | 1 | 0 | 1
  Skin: Abnormal at BL → Normal at EP | 0 | 1 | 0 | 1
  Skin: Abnormal at BL → Abnormal at EP | 3 | 3 | 3 | 1
  Lymph Nodes: Normal at BL → Normal at EP | 25 | 26 | 24 | 27
  Lymph Nodes: Normal at BL → Abnormal at EP | 0 | 1 | 0 | 0
  Lymph Nodes: Abnormal at BL → Normal at EP | 0 | 0 | 1 | 0
  Lymph Nodes: Abnormal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  Neurological: Normal at BL → Normal at EP | 26 | 28 | 27 | 27
  Neurological: Normal at BL → Abnormal at EP | 0 | 0 | 0 | 0
  Neurological: Abnormal at BL → Normal at EP | 0 | 1 | 0 | 0
  Neurological: Abnormal at BL → Abnormal at EP | 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through Week 12
Arm/Group | Placebo | Armodafinil 50 mg/Day | Armodafinil 150 mg/Day | Armodafinil 250 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 14/29 | 15/30 | 16/29 | 16/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Armodafinil 50 mg/Day (N=30) | Armodafinil 150 mg/Day (N=29) | Armodafinil 250 mg/Day (N=29)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 5 | 5 | 5
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 4 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 3 | 1
Bruxism (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Initial insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Logorrhoea (Psychiatric disorders) | 0 | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Tachyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0
Pressure of speech (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The sponsor's decision to terminate the study early resulted in a small number of study participants and related limitations to the interpretation of the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.